CLINICAL TRIAL: NCT04101435
Title: Immunogenicity and Safety Evaluation of AdimFlu-S Quadrivalent Inactivated Influenza Vaccine (QIS) in Healthy Subjects Aged 3 Years Old to 17 Years Old
Brief Title: Immunogenicity and Safety Evaluation of QIS in Healthy Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adimmune Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ADIMQIS20160328
Record Dates: First submitted 2019-09-17; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Influenza
Keywords: Influenza Vaccine; Immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Aged 3 to 8 years old vaccine naïve subject (without prior seasonal influenza vaccine exposure)
  Interventions: Biological: AdimFlu-S (QIS)
- Group B (Active Comparator): Aged 3 to 8 years old vaccine non-naïve subject (with prior seasonal influenza vaccine exposure)
  Interventions: Biological: AdimFlu-S (QIS)
- Group C (Experimental): Aged 9 to 17 years old subject
  Interventions: Biological: AdimFlu-S (QIS)

INTERVENTIONS:
Biological: AdimFlu-S (QIS) — This was an open study to demonstrate the use of AdimFlu-S (QIS) (2016-2017 season) vaccine in young subjects aged between 3 years old to 17 years old. All subjects were divided into two subgroups. That were subjects aged 3 to 8 years old, who received 2 doses of 0.5 mL vaccine separated by 4 weeks, and subjects aged 9 to 17 years old, who received one dose of 0.5 mL vaccine.

SUMMARY:
The purpose of this study was to evaluate the antibody response to each of the four influenza vaccine strains included in the study vaccine, as measured by hemagglutination inhibition (HAI) at 4 weeks after the last dose of the study vaccine in young subjects aged between 3 years old and 17 years old.

ELIGIBILITY:
Inclusion Criteria:

1. Boys or girls aged 3 years old to 17 years old on the day of first vaccination;
2. Subject and/or parents(s)/legal guardian(s) must be willing to comply with planned study procedures and be available for all study visits;
3. Subject must be in good physical health on the basis of medical history, physical examination;
4. Subject and/or parents(s)/legal guardian(s) must read and signed the study-specific informed consent prior to initiation of any study procedure.

Exclusion Criteria:

Main exclusion criteria:

1. Subjects received influenza vaccine (Trivalent and/or Quadrivalent) within 6 months prior first vaccination.
2. History of hypersensitivity to eggs or egg protein or similar pharmacological effects to study medication;
3. Personal or family history of Guillain-Barré Syndrome;
4. An acute febrile illness within 1 week prior to vaccination;
5. Current upper respiratory illness (URI), including the common cold or nasal congestion within 72 hours prior to vaccination;
6. Subjects with influenza-like illness as defined by the presence of fever (temperature >38ºC) and at least two of the following four symptoms: headache, muscle/joint aches and pains (e.g. myalgia/arthralgia), sore throat and cough;
7. Female subjects who were pregnant, lactating or likely to become pregnant during the study; Women of childbearing potential disagreed to use an acceptable method of contraception (e.g., hormonal contraceptives, IUD, barrier device or abstinence) throughout the study;
8. Treatment with an investigational drug or device, or participation in a clinical study, within 3 months before consent;
9. Immunodeficiency, or under immunosuppressive therapies;
10. Receipt of live virus vaccine within 1 month prior to study vaccination or expected to receive vaccination before the last blood sampling for immunogenicity evaluation;
11. Receipt of any inactivated vaccine within 2 weeks prior to study vaccination or expected to receive vaccination before the last blood sampling for immunogenicity evaluation;
12. Receipt of any blood products, including immunoglobulin from 3 months before first vaccination to the last blood sampling for immunogenicity evaluation;
13. Underlying condition in the investigators' opinion might interfere with evaluation of the vaccine.

3. Treatment discontinuation

1. Withdrawal criteria i. Subject/Subject's guardians decided to withdraw consent. ii. Lost to follow-up. iii. Administration of prohibited medication/treatment/vaccine. iv. Any pathological event, clinical adverse event, or any change in the subject's status giving indication to the pediatrician that further participation in the study might not be the best interests of the subject, according to investigator's discretion.
2. Contraindications to second vaccination

Subject with any of the following criteria might be contraindicated to take the second vaccination:

i. Had any Grade 3 or Grade 4 adverse reaction within 7 days after first dose. ii. Had any SAE related to first dose during the follow-up of first dose. iii. Any situations met the exclusion criteria, except the exclusion criterion (1) and (8).

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 174 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2017-07-12 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
Evaluate the immunogenicity profiles for influenza virus vaccine strains of the AdimFlu-S (QIS) by seroconversion rate | Change from baseline for anti-hemaglutinin antibodies at 28 days post immunization
  The primary endpoint of immunogenicity evaluation was the seroconversion rate
Evaluate the immunogenicity profiles for influenza virus vaccine strains of the AdimFlu-S (QIS) by geometric mean folds increase | Change from baseline for anti-hemaglutinin antibodies at 28 days post immunization
  The primary endpoint of immunogenicity evaluation was the geometric mean folds increase

SECONDARY OUTCOMES:
Evaluate the immunogenicity profiles for influenza virus vaccine strains of the AdimFlu-S (QIS) by seroprotection rate | Change from baseline for anti-hemaglutinin antibodies at 28 days post immunization
  The secondary endpoint of immunogenicity evaluation was the seroprotection rate
Evaluate the safety and tolerability profiles including the presence or absence of the pre-specified reactogenicity events and other serious/non-serious adverse events of the AdimFlu-S (QIS) | In regard to the long term safety of the study vaccine, the significant and/or serious adverse event(s) will be recorded during the 6 months follow up after the scheduled last vaccination
  Evaluate the safety and tolerability profiles including the presence or absence of the pre-specified reactogenicity events and other serious/non-serious adverse events of QIS. Reactogenicity events were pre-specified adverse events systematically recorded on diary cards during post-vaccination period by all participants for 7 days after each vaccination. Unsolicited adverse events were recorded on the diary card till 28 days post vaccination, while serious adverse events should be recorded throughout the study period

IPD SHARING:
Plan to Share IPD: No